CLINICAL TRIAL: NCT01760330
Title: A Prospective, Double-Blinded, Randomized Comparison of Intravenous Acetaminophen Versus Placebo in Children Undergoing Palatoplasty
Brief Title: IV Acetaminophen in Children Undergoing Palatoplasty
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to obtain funding
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Tarun Bhalla, MD, Clinical Assistant Professor, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB12-00709
Record Dates: First submitted 2012-12-12; First posted 2013-01-04 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Cleft Palate
MeSH Terms: conditions — Cleft Palate | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IV acetaminophen (Active Comparator): IV acetaminophen administered q 4 hrs. for a total of 24 hrs.
  Interventions: Drug: IV acetaminophen
- Placebo (Placebo Comparator): Normal saline administered IV every 4 hrs. for a total of 24 hrs.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IV acetaminophen
  Other Names: Ofirmev
  Arms: IV acetaminophen
Drug: Placebo
  Arms: Placebo

SUMMARY:
This project is being used to assess the utility of intravenous acetaminophen in the pediatric population undergoing palate repairs. This study is a prospective randomized double blinded placebo controlled study. The investigators will have two arms, one group of patients will receive intravenous acetaminophen and one group that will receive a placebo at a total of four doses over 24 hours. The results of this study may affect the intraoperative anesthetic management as well as post-operative surgical management of this specific patient population. The goal is to determine the benefit of adding a non-opioid analgesic and hypothesizing that it may reduce the amount of narcotic consumption in the post anesthesia care unit as well as during the post-operative stay.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I or II
* Presenting for repair of palatoplasty with Drs. Kirschner or Pearson

Exclusion Criteria:

* ASA physical status > II
* Underlying Syndrome
* Significant co-morbid diseases (cardiac, pulmonary, neurological disease)
* Patients having concomitant procedures (tonsillectomy, adenoidectomy, etc.)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Pain | 24 hrs. post-op.
  Pain scores will be assessed.

SECONDARY OUTCOMES:
Opioid consumption | 24 hrs. post-op

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States